CLINICAL TRIAL: NCT01176890
Title: The Significance of Intact Vagal Innervation for the GLP-1 Induced Inhibition of Gastric Emptying, Appetite and Food Intake
Brief Title: Intact Vagal Innervation and Glucagon-like Peptide-1 (GLP-1) Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jonatan I Bagger, MD, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Truncated mealtest (AP)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Vagotomy, Truncal
Keywords: truncal vagotomy; GLP-1; gastric emptying; appetite; food intake
MeSH Terms: interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vago (Experimental): Truncally vagotomized subjects (due to duodenal ulcer operation)
  Interventions: Drug: GLP-1; Other: Saline
- Cardia (Experimental): truncally vagotomized subjects (due to esophagus resection)
  Interventions: Drug: GLP-1; Other: Saline
- Healthy controls (Experimental): Healthy control subjects
  Interventions: Drug: GLP-1; Other: Saline

INTERVENTIONS:
Drug: GLP-1 — 1.2 pmol/kg/min GLP-1 will be infused intravenously during the four hour meal test (100 g Ny NAN1 and 1.5 g paracetamol dissolved in 300 ml water) ingested over 10 minutes.
  After four hours an ad libitum meal will be supplied
  Other Names: Panodil
Other: Saline — Saline (isotonic NaCl) will be infused intravenously during the four hour meal test (100 g Ny NAN1 and 1.5 g paracetamol dissolved in 300 ml water) ingested over 10 minutes.
  After four hours an ad libitum meal will be supplied
  Other Names: Panodil

SUMMARY:
The aim of this study is to investigate the role of transmission via the vagal nerve for the effect of Glucagon-like peptide-1 (GLP-1) in respect to gastric emptying, appetite and food intake.

The hypothesis is that a great deal of the effects of GLP-1 is mediated via the nervous system and for this reason the researchers will investigate individuals with and without intact nervous supply.

DETAILED DESCRIPTION:
GLP-1 is a potent enterogastron and incretin hormone. It is rapidly inactivated by dipeptidyl peptidase IV so only 10-15% enters the systemic circulation. This has led to the hypothesis that GLP-1 interact locally with afferent sensory nerve fibers. We investigated the role of intact vagal innervations on the effect of GLP-1 on the food intake, gastric emptying (GE) and appetite.

ELIGIBILITY:
Inclusion Criteria:

* truncal vagotomy
* normal hemoglobin
* informed consent
* Age, gender and weight matched controls
* normal hemoglobin
* informed consent

Exclusion Criteria:

* type 1 diabetes mellitus or type 2 diabetes mellitus
* body mass index > 30 kg/m2
* inflammatory bowel disease
* intestinal resection
* nephropathy (serum creatinine > 150 µM and/or albuminuria)
* liver disease (ALAT and/or ASAT > 2 x normal value)
* treatment with medicine which cannot be paused for 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Gastric emptying | four hours
  Gastric emptying will be assessed using a liquid meal with 1.5 g paracetamol added and continuous blood sampling for measuring paracetamol concentration during four hours
Appetite | four hours
  Hunger, satiation, and fullness will be assessed before, during and after a liquid meal with 1.5 g paracetamol added using a visual analog scale (VAS)
Food intake | five hours
  After the liquid meal test, the volunteers will be offered a meal to assessed their ad libitum food intake

SECONDARY OUTCOMES:
plasma glucose | four hours
serum insulin and c-peptide | four hours
plasma glucagon | four hours
plasma GLP-1 | four hours
endogenous GLP-1 | four hours
  endogenous GLP-1 will be assessed as plasma GLP-2 concentration
plasma GIP | four hours
serum paracetamol | four hours

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Plamboeck, M.D., Principal Investigator — University Hospital, Gentofte, Copenhagen; Tina Vilsbøll, M.D., Study Director — University Hospital, Gentofte, Copenhagen
Locations (1):
- Department of Internal Medicine F' laboratory, Hellerup, Copenhagen, Denmark

REFERENCES:
- [Derived] Wewer Albrechtsen NJ, Hartmann B, Veedfald S, Windelov JA, Plamboeck A, Bojsen-Moller KN, Idorn T, Feldt-Rasmussen B, Knop FK, Vilsboll T, Madsbad S, Deacon CF, Holst JJ. Hyperglucagonaemia analysed by glucagon sandwich ELISA: nonspecific interference or truly elevated levels? Diabetologia. 2014 Sep;57(9):1919-26. doi: 10.1007/s00125-014-3283-z. Epub 2014 Jun 3. PMID 24891019
- [Derived] Plamboeck A, Veedfald S, Deacon CF, Hartmann B, Wettergren A, Svendsen LB, Meisner S, Hovendal C, Vilsboll T, Knop FK, Holst JJ. The effect of exogenous GLP-1 on food intake is lost in male truncally vagotomized subjects with pyloroplasty. Am J Physiol Gastrointest Liver Physiol. 2013 Jun 15;304(12):G1117-27. doi: 10.1152/ajpgi.00035.2013. Epub 2013 Apr 18. PMID 23599045